CLINICAL TRIAL: NCT04184973
Title: Efficacy and Safety of the CG-100 Intraluminal Bypass Device in Colorectal and Coloanal Anastomoses: Prospective, Open Label, Randomized Trial
Brief Title: Efficacy and Safety of the CG-100 Intraluminal Bypass Device
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Colospan Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CLD-075
Record Dates: First submitted 2019-12-01; First posted 2019-12-04 (Actual); Last update posted 2025-10-23 (Actual); Status verified 2025-10

CONDITIONS: Rectal Cancer; Rectal Tumor; Rectal/Anal
Keywords: anastomosis; leak; mesorectal; ileostomy; colostomy
MeSH Terms: conditions — Rectal Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- CG-100 (Experimental): Patients receive CG-100 during rectal cancer surgery
  Interventions: Device: CG-100 intraluminal bypass device
- SOC (Active Comparator): Patients receive a protective stoma during rectal cancer surgery
  Interventions: Procedure: Stoma

INTERVENTIONS:
Device: CG-100 intraluminal bypass device — a removable, temporary intraluminal bypass device, developed by Colospan, is designed to safely postpone the creation of a protective stoma until 10 days after surgery only for patients who need it (i.e. have a defect in the anastomosis)
  Arms: CG-100
Procedure: Stoma — Primary protective ileostomy
  Arms: SOC

SUMMARY:
A randomized trial to assess the safety and efficacy of CG-100 for reducing stoma creation rate in subjects undergoing mesorectal excision.

DETAILED DESCRIPTION:
A primary diverting stoma is widely used by surgeons in order to bypass the low rectal anastomosis and reduce morbidity associated with anastomotic leaks. Today a stoma is created for all high-risk patients even though the expected anastomotic leak rate is less than 20%. This means that 80% of patients are exposed to potentially serious complications associated with the stoma itself without any clinical benefit.

CG-100, a removable, temporary intraluminal bypass device, developed by Colospan, is designed to address this need by safely postponing the creation of a protective stoma until 10 days after surgery only for patients who need it (i.e. have a defect in the anastomosis); thereby allowing patients with an intact anastomosis a quicker and safer return to normal activity.

ELIGIBILITY:
Inclusion Criteria:

1. The patient is willing to comply with protocol-specified follow-up evaluations
2. Patient 22-65 years of age at screening, or patient 66-70 years of age at screening with up to one cardiovascular, metabolic or pulmonary comorbidity for which medication is prescribed.
3. Patient is diagnosed with colorectal cancer
4. Patient is scheduled for elective either open, laparoscopic or robotic with mesorectal excision (either abdominal or transanal approach) which will require the creation of an anastomosis, maximally 10 cm from the anal verge
5. Patients who are scheduled to receive a protective stoma under routine clinical practice during their primary planned operation.
6. Patient is scheduled to undergo mechanical bowel preparation
7. The patient has been informed of the nature of the study, agrees to its provisions and has provided written informed consent, approved by the appropriate Medical Ethics Committee (EC) or Institutional Review Board (IRB).

Exclusion Criteria:

1. Patient has local or systemic infection at the time of intervention (e.g., peritonitis)
2. Major surgical or interventional procedures within 45 days prior to this study or planned surgical or interventional procedures within 6 months of entry into this study (not including, placement of port for chemotherapy or ureter stent insertion).
3. Patients with ASA classification > 3
4. Albumin < 30 g/liter
5. Patient has a diagnosis of bowel obstruction, bowel strangulation, peritonitis, bowel perforation, ischemic bowel, carcinomatosis or extensively spread inflammatory bowel disease
6. Patients has a diagnosis of coagulopathy, thrombocytopenia, immune suppression
7. BMI ≥ 40
8. Patient is going through another surgical procedure (other than ileostomy, adhesiolysis) during the surgery.
9. The patient is currently participating in another investigational drug or device study unless pre-approved by the sponsor.
10. Patient has been taking regular systemic/ steroid medication in the last 6 months.
11. Patients is taking antimetabolites or antiplatelet agents.
12. Patient has preexisting sphincter problems
13. Patient has evidence of extensive local disease in the pelvis or has undergone a prior pelvic anastomosis.
14. Patients with massive diverticulosis at the sigmoid/descending colon (viewed on preoperative CT)
15. Any condition or abnormality which in the opinion of the investigator may jeopardize the patient's safe participation or the quality of the data
16. Pregnant or nursing female patients. Female patients of child-bearing potential must have a negative pregnancy test done within 7 days prior to surgical procedure per site standard test.

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Estimated)
Dates: Start 2020-06-23 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in Stoma creation rate | 39 Weeks
Incidence of complications | 39 Weeks

CONTACTS AND LOCATIONS:
Locations (14):
- United States (10):
  - University of California Irvine, Orange, California
  - Kaiser Permanente San Diego medical Center, San Diego, California
  - Colorado University Anschutz Medical Campus, Aurora, Colorado
  - University of Louisville, Louisville, Kentucky
  - Henry Ford Health System, Detroit, Michigan
  - East Bank Hospital - M Health Fairview University of Minnesota Medical Center, Minneapolis, Minnesota
  - New York-Presbyterian / Weill Cornell Medical Center, New York, New York
  - Jefferson University Hospital, Philadelphia, Pennsylvania
  - Lifespan & Brown Surgical Associates, Providence, Rhode Island
  - University of Utah Health, Salt Lake City, Utah
- Israel (3):
  - Soroka University Medical Center, Beersheba
  - Carmel Medical Center, Haifa
  - Rabin Medical Center, Petah Tikva
- Humanitas Research Hospital, Milan, Lombardy, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: U.S. Clinical Study Website — https://stomachoice.com/